CLINICAL TRIAL: NCT06693180
Title: Registry Hyperbaric Oxygen in Diabetic Foot Ulcer
Brief Title: Registry HBOT in DFU
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, Dirk T. Ubbink, Prof., University of Amsterdam
Other Study IDs: 2024.0066
Record Dates: First submitted 2024-11-07; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Diabetic Foot Ulcers
Keywords: HBOT; Diabetic foot ulcer; Hyperbaric Oxygen Therapy; DFU; Peripheral arterial disease
MeSH Terms: conditions — Diabetic Foot; Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- HBOT: Received complementary HBOT
  Interventions: Other: HBOT
- Control: Standard care therapy

INTERVENTIONS:
Other: HBOT — Hyperbaric Oxygen Therapy
  Groups: HBOT

SUMMARY:
Overview of available data to assess the benefits of HBOT to DFU patients

DETAILED DESCRIPTION:
10 year retrospective registry to measure outcomes regarding major amputations, mortality, hospital admissions in patients with a diabetic foot ulcer with peripheral ischaemia. Two groups will be compared: complementary HBOT and a control group.

ELIGIBILITY:
Inclusion Criteria:

* Diabetes mellitus
* Meggitt-Wagner classification grade 2-4, existing > 4 weeks
* Complete 1 year follow-up

Exclusion Criteria:

* Chronic Obstructive Pulmonary Disease (COPD) GOLD IV
* Treatment with chemotherapy, immunosuppressive drugs or systemic corticosteroids within the last 3 months
* Metastasized malignancy
* Left ventricular ejection fraction (EF) <20% or external pacemaker
* Recent thoracic or middle ear surgery
* Severe epilepsy
* Uncontrollable high fever
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients suffering from diabetes and peripheral ischaemia who have a diabetic foot ulcer for longer than 4 weeks.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Major amputation rate | 1 year
  Major (above the ankle) amputation rate

SECONDARY OUTCOMES:
Mortality | 1 year
  Mortality
Amputation-free survival rate | 1 year
  Amputation-free survival rate: percentage of patients who are alive with their leg.
Complete wound healing | 1 year
  Complete wound healing
Pain score | 1 year
  Pain score (10-point Visual Analogue Scale; 0= no pain, 10 is intolerable pain)
Additional vascular interventions | 1 year
  Additional vascular interventions

CONTACTS AND LOCATIONS:
Overall Officials: Joost R Meijering, MD, Study Chair — Amsterdam University Medical Center; Dirk T Ubbink, MD, PhD, Principal Investigator — Amsterdam University Medical Center
Locations (1):
- Amsterdam UMC, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No